CLINICAL TRIAL: NCT02859688
Title: Can Epimutations be Inherited? How to Manage Patients With Imprinting-related Diseases Who Wish to Become Parents
Acronym: REPAR
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: BRUNO AOI 2014
Record Dates: First submitted 2016-08-02; First posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-07

CONDITIONS: Epimutation
MeSH Terms: interventions — High-Throughput Nucleotide Sequencing; Epigenome

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, sperm, saliva, skin biopsy

GROUPS / COHORTS (3):
- SRS patient
  Interventions: Genetic: pyrosequencing; Genetic: Methylome
- father SRS patient
  Interventions: Genetic: pyrosequencing; Genetic: Methylome
- control patient
  Interventions: Genetic: pyrosequencing; Genetic: Methylome

INTERVENTIONS:
Genetic: pyrosequencing
Genetic: Methylome

SUMMARY:
Like genetic mutations, DNA methylation anomalies or epimutations can disrupt gene expression and lead to human diseases.

However, unlike genetic mutations, epimutations can in theory be reverted through developmental epigenetic re-programing, which should limit their transmission across generations. Following the request for a parental project of a patient diagnosed with Silver-Russell syndrome (SRS), and the availability of both somatic and spermatozoa DNA from the proband and his father, we had the exceptional opportunity to evaluate the question of inheritance of an epimutation. We provide here for the first time evidence for efficient reversion of a constitutive epimutation in the spermatozoa of an SRS patient, which has important implication for genetic counseling.

ELIGIBILITY:
Inclusion Criteria:

* Men who have been informed about the study
* Patients over 18 years old
* Fertile
* Matched for age with Silver Russel syndrome (SRS) patients

Exclusion Criteria:

* Adults under guardianship
* Patients without national health insurance cover
* Patients with psychomotor development diseases or pulmonary, cardiac, renal or metabolic diseases (including type 1 and 2 diabetes before the pregnancy), inflammatory and systemic diseases, hypertension, neurological diseases, chronic hepatitis B or C, infection with human immunodeficiency virus (HIV).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1 patient SRS, the father of the patient SRS and 5 control patients : healthy men, age-matched
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Analysis of levels of methylation of deoxyribonucleic acid (DNA) measured by cloning/ sequencing and/or pyrosequencing for genes susceptible to imprinting (GSI) | Through the study completion up to 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France